## Integrated Alcohol Disorder and PTSD Treatment

NCT01601067

04/14/2016

## Objectives

The primary aim will be to evaluate the effects on alcohol use and PTSD symptoms of an exposure-based integrated AD and PTSD intervention (i.e., COPE) when compared to a present-focused coping skills intervention (i.e., Seeking Safety [SS]) in male and female Veterans with comorbid AD and PTSD. Hypotheses for the primary aim are:

- 1. At post-treatment, both groups will show reductions in alcohol use, but COPE will demonstrate greater reduction in PTSD symptoms than SS.
- 2. At the 2nd and 3rd post treatment follow up assessment ,COPE will have significantly fewer percent drinking days than SS.
- 3. At the 2nd and 3rd post treatment follow up assessment ,COPE will continue to have lower PTSD symptom scores.

## Design.

The proposed study will be a randomized controlled trial comparing. Concurrent Treatment of PTSD and Substance Use Disorders using PTSD (COPE) to Seeking Safety (SS) for the treatment of male and female Veterans with AD/PTSD. 178 participants will be enrolled through the San Diego VA and randomized at the individual level. Measures will occur at baseline, post-treatment, and two post treatment follow up assessments. Participants will complete the 2nd post treatment assessment interview and set of questionnaires 3 months after the 1st post treatment appointment. Participants will be scheduled for their 3<sup>rd</sup> and last post treatment interview 3 months after completing their 2<sup>nd</sup> post treatment assessment. All procedures will be done for research purposes.

## Methods

All work will be carried out at the SAMI outpatient program and PTSD clinics of the Veteran Affairs San Diego Healthcare Systems (VASDHS). Random permuted blocks will be used which ensure exactly equal treatment numbers at certain equally spaced points in the sequence of patient assignment. Randomization will be stratified by gender to ensure a balanced number of males and females are in each treatment group.

The <u>Timeline Follow-back Procedure (TLFB50)</u> will be employed at baseline, post-treatment, 5-month, and 8-month follow up to evaluate drinking and all drug use during the 30 days preceding each interview.

The <u>Clinician-Administered PTSD Scale for DSM-V(CAPS54,55)</u> is a standard semi-structured interview used to assess PTSD diagnosis and severity. As part of the CAPS, a list of potentially traumatic events is given to respondents.

Eligible participants will contact our study in response to flyers/ brochures posted in San Diego VA hospital, including the Mission Valley, Chula Vista, and Oceanside CBOCS; and by referral from VA primary care, substance use mental illness (SAMI), PTSD (OEF/OIF/OND, PCT, MST), and other clinics (ADTP, SARRTP); and also from VASDHS and VMRF websites under "Research opportunities"